CLINICAL TRIAL: NCT02036944
Title: Celiac Disease and Unexplained Iron Deficiency in a Primary Care Setting
Status: Terminated | Type: Observational
Why Stopped: Study stopped d/t lack of enrollment and no compelling data.
Sponsor: Providence Medical Research Center (Other)
Collaborators: Providence Sacred Heart Medical Center & Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMRC-1909-1
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Celiac Disease; Iron Deficiency; Iron Malabsorption
Keywords: Celiac Disease; Celiac Sprue; Iron-Deficiency Anemia
MeSH Terms: conditions — Celiac Disease; Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — The serum remaining from 10 mL of blood will be aliquoted and frozen at -70 degrees. If future funding allows, these samples will be tested for autoimmune and malabsorption markers.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if patients with unexplained iron deficiency have underlying diseases processes such as celiac disease.

It is hypothesized that selectively screening patients with unexplained iron deficiency will reveal previously undiagnosed etiologies, including celiac disease and other causes of iron malabsorption along with various sources of occult GI blood loss.

DETAILED DESCRIPTION:
The primary purpose of the study is to document unexplained iron deficiency and its relationship to celiac disease, iron malabsorption and occult intestinal blood loss. Test results given to primary care physicians may prompt further testing for celiac disease (duodenal biopsy) or other potential causes of occult iron deficiency. The specific endpoints to be evaluated include:

* Prevalence of specific serum markers of celiac disease in those with unexplained serum markers of iron deficiency.
* Prevalence of iron malabsorption with and without celiac disease in the same population
* Frequency of other blood tests for malabsorption and their association with celiac disease or other cause of iron malabsorption.
* Frequency of specific historical markers associated with celiac disease
* Prevalence of unrecognized GI blood loss
* Quality of life improvement based on new diagnoses with appropriate therapy
* After one year follow-up, review patient records for additional diagnoses explaining iron deficiency.

Primary Objective:

Discover several etiologies of unexplained iron deficiency in a primary care clinic population including celiac disease, iron malabsorption and occult intestinal blood loss.

Secondary Objectives:

* Define percent of total clinic patient population with one or more markers of iron deficiency on last testing and the subset without an apparent etiology on their problem list ("study group").
* Define percent of patients in the study group that are currently iron deficient at time of study onset, and how many of those are actually anemic.
* Define percent of study group patients with iron malabsorption, with or without celiac disease.
* Document improved quality of life outcomes for those with new diagnoses and appropriate therapy, including celiac disease given gluten-free diet and iron therapy.
* For those patients identified with celiac disease, do statistical analysis of historical and lab parameters that are more highly linked to celiac disease to improve screening parameters.
* Document percent of various diagnoses that explain occult iron deficiency as found by primary care providers over the course of a one year follow-up after initial diagnosis. (Providers will be given all testing results related to their patients after the initial screening and at one year.)
* Specific cost-effectiveness of this screening procedure may be done in a future study if preliminary results are suggestive of improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Active outpatients in the Providence Internal Medicine Residency Clinic, Family Medicine Residency Clinics, or Providence Internal Medicine Clinic
2. Demographic Age > 18 years. Diagnostic criteria: markers of iron deficiency at last check are defined as MCV<80 fL, Iron Sat<20% or ferritin<30 ng/mL.
3. Patient signs informed consent document and HIPAA authorization for release of personal health information.
4. Ability to understand procedures and comply with them for one year duration of study

Exclusion Criteria:

1. Any documented significant acute or chronic blood loss, per medical record review or self- report (see Appendix B). Significant blood loss includes

   1. Acute blood loss requiring iron treatment or transfusions within 1 year prior to the above measure of iron deficiency
   2. Chronic blood loss (such as menorrhagia, GI bleeding, hemoptysis, hematuria, chronic nose bleeds, hemolysis, regular blood donations, or major trauma requiring transfusion or iron therapy)
   3. Thalassemia or other major hemolytic diseases.
2. Prior diagnosis of celiac disease, or other documented cause of iron malabsorption.
3. Women who are currently pregnant, or who were pregnant with 6 months prior to time of last testing.
4. Those currently or recently on chemotherapy (within the last 6 months)
5. Those with prior gastric resection or bariatric surgery
6. Those with advanced chronic kidney disease (stage 4 or 5)
7. Any other reasons that, in the investigators' opinion, may prevent compliance with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Providence Internal Medicine Clinic, Providence Internal Medicine Residency Services and Providence Family Medicine Residency Services
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Positive results for Expanded Celiac Disease Panel | Upon consent and enrollment in the study, laboratory tests will be done to evaluate for the presence of Celiac Disease
  Expanded Celiac Disease Panel includes TTG-IgG, TTG-IgA, AntiGliadin-IgG, AngtiGliadin-IgA, and Total Serum IgA

SECONDARY OUTCOMES:
Percentage of Clinic Patient Population with one or more markers of iron deficiency | at enrollment
  Other tests will be done at enrollment to assess for iron malabsorption and possibly to identify causes of iron malabsorption other than celiac disease. These include Iron absorption Testing (serum iron level before and after oral FeSO4 tablet or liquid), with percent iron saturation. Ferritin, Hemoglobin and Hematocrit, Vitamin D level, Folate, Vitamin B12 level, Aspartate Aminotransferase (AST), and Stool Occult Blood Test

OTHER OUTCOMES:
Improved Quality of Life after one year of intervention (either gluten-free diet if Celiac disease is diagnosed and/or recommendation of daily iron supplementation) | Enrollment and End of One Year
  For patients diagnosed with Celiac disease at enrollment, a gluten-free diet will be advised explained by a Registered Dietician. Patients not diagnosed with celiac disease but with iron deficiency or malabsorption will be advised to take daily oral iron supplements. Quality of Life Surveys will be administered at enrollment and at the end of one year to assess for improvement resulting from diet and/or supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Palpant, MD, Principal Investigator — Providence Internal Medicine Residency Services
Locations (1):
- Providence Medical Research Center, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No